CLINICAL TRIAL: NCT06149884
Title: Micrometastases in Axillary Lymph Nodes in Breast Cancer, Post-neoadjuvant Chemotherapy
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Joon Jeong, Proffesor, Gangnam Severance Hospital
Other Study IDs: 3-2023-0214
Record Dates: First submitted 2023-11-14; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Micrometastases; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Neoplasm Micrometastasis | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sentinel lymph node biopsy, axillary lymph node dissection — SLNB was performed using single or dual tracers. For the single tracer technique, Technetium 99, a radioactive substance, was administered periareolarly prior to surgery, and SLNs were identified intraoperatively via a gamma detection system (Neoprobe®). The dual tracer method employed both an isosulfan blue dye and Technetium 99 concurrently. The choice of SLNB technique was contingent upon the surgeon's discretion. SLNs were categorized as one or multiple, and any LN identified by either or both methods was defined as SLN. LNs resected during SLNB without tracer signal were not classified as SLNs.
  ALND was characterized by the removal of all LNs in axillary levels I and II. Patients documented to have undergone ALND in surgical records were primarily selected from our registry. Among them, those with fewer than 10 LNs were excluded, based on the assumption that a competent ALND necessitated the removal of 10 or more LNs as defined in previous studies

SUMMARY:
This study aims to investigate the significance of minimal residual axillary disease following NAC, with a particular focus on micrometastases (ypNmi), in comparison to pathologic lymph node-negative (ypN0) or macrometastases (ypN+). The investigators will further explore the prognostic implications of SLNmi for the prediction of axillary LN status and survival outcomes.

DETAILED DESCRIPTION:
This study aims to investigate the significance of minimal residual axillary disease following NAC, with a particular focus on micrometastases (ypNmi), in comparison to pathologic lymph node-negative (ypN0) or macrometastases (ypN+). The investigators will further explore the prognostic implications of SLNmi for the prediction of axillary LN status and survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Stage II or III primary breast cancer patients
* Patients who performed neoadjuvant chemotherpay
* Patients who underwent axillary lymph node dissection with or without sentinel lymph node biopsy

Exclusion Criteria:

* Patients who performed upfront surgery
* De novo stage IV patients

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We conducted a retrospective review of primary breast cancer patients from the breast cancer registries of Gangnam Severance Hospital and Severance Hospital, who underwent surgery following NAC between September 2006 and February 2018. These patients were clinically diagnosed with stage II or III breast cancer and underwent ALND, with or without SLNB. The surgical approach, encompassing either total mastectomy or breast-conserving surgery, was dictated by the number and size of the tumors present. Exclusion criteria comprised of patients who had initial surgery, underwent only SLNB, or presented with de novo stage IV disease.
Sampling Method: Non-Probability Sample
Enrollment: 978 (Actual)
Dates: Start 2006-09-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival | the interval from breast cancer diagnosis to the initial recurrence or death upto 5 years
  locoregional recurrence, distant metastasis, any cause of death